CLINICAL TRIAL: NCT03394391
Title: A Single-blind, Randomized, Parallel Design Study to Assess the Effectiveness of SMS Reminders in Improving ART Adherence Among Adolescents Living With HIV in Nigeria (STARTA Trial-Adolescents)
Brief Title: The Effectiveness of SMS in Improving Antiretroviral Medication Adherence Among Adolescents Living With HIV in Nigeria
Acronym: STARTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Olumide ABIODUN (Other)
Responsible Party: Sponsor-Investigator, Dr. Olumide ABIODUN, Senior Lecturer and Honorary Consultant, Babcock University
Organization: Babcock University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: BUTH/CT/0001; MISP Database number #57473 (Other Grant/Funding Number: MERCK SHARP & DOHME CORP.)
Record Dates: First submitted 2017-12-28; First posted 2018-01-09 (Actual); Results first posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: HIV Infections
Keywords: Adherence; Adolescents; Antiretroviral therapy; HIV; Nigeria; Randomized controlled trial; Short message services
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: A single-blind, parallel-design (ratio 1:1), and multi-centre RCT of 230 adolescent living with HIV who are non-adherent to medications will be conducted over a one-year period in Southwest Nigeria.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators, data manager, research assistants, counselors and other project staff will be blinded throughout the study. An independent medical internet technology firm will be contracted to randomize participants and to send the required SMS to the participants. After scientific review has been completed and data collection has been completed, at the point of analysis, a list of participants' unique identifiers in two groups will be sent to the data analysts without specifying which the investigation or control group is. The blinding of the clinical database will finally be removed after final data analysis has been completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Daily ART-adherence SMS reminder
  Interventions: Behavioral: Daily ART-adherence SMS reminder; Behavioral: Standard Adherence Counselling/Patient experience group chat
- Control group (Active Comparator): Standard adherence counselling/Patient experience group chat
  Interventions: Behavioral: Standard Adherence Counselling/Patient experience group chat

INTERVENTIONS:
Behavioral: Daily ART-adherence SMS reminder — Interactive and tailored SMS reminders that are acceptable to the participants to remind them to take their medications and to make clinic attendance.
  Arms: Intervention group
Behavioral: Standard Adherence Counselling/Patient experience group chat — All the participants will receive the standard adherence counselling by trained counsellors at each visit.
  All participants will also be enlisted in a group chat on social media where they will discuss their experiences with the quality of HIV services rendered at their respective clinics. A specialist who will have very minimal involvement will give weekly feedback and counsel on how best to resolve prominent challenges.

SUMMARY:
The non-maintenance of ART adherence is a major barrier to the achievement of optimal treatment outcomes among adolescents living with HIV. ART adherence is a challenge among adolescents living with HIV because of lack of appropriate information, their unique emotional state and lifestyles but the most commonly quoted challenge to adherence is forgetting to take antiretroviral drugs. There is evidence to suggest that short message service (SMS) reminder- interventions may enhance drug compliance among adolescents living with other chronic diseases such as asthma and diabetes. Available literature underscores the need for randomized controlled trials (RCTs) of effective interventions to promote ART adherence among adolescents with HIV.

The aim of this study is to evaluate the feasibility, acceptability, and efficacy of interactive and tailored SMS reminders on ART adherence among adolescents (15-19 years) living with HIV in Ogun State, Nigeria. The study hypothesizes that the use of personal mobile phones and SMS reminders for the improvement of ART adherence among adolescents living with HIV are feasible, acceptable, and effective.

A single-blind, parallel-design (ratio 1:1), and multi-center RCT of 230 adolescent living with HIV who are non-adherent to medications will be conducted over a one-year period in Southwest Nigeria. All the participants will receive routine adherence counseling during clinic visits and one SMS reminder each for follow-up appointments 48 hours and 24 hours before the follow-up visit date. The intervention group will also receive daily ART adherence reminder SMS. Participants will be assessed at baseline and during follow-up visits at 4, 8, 12, 16 and 20 weeks after the baseline. Baseline assessment of participants will include socio-demographic characteristics; HIV/AIDS risk behaviour assessment, Alcohol and Drug abuse assessment, Client Satisfaction Survey, ART adherence assessment, CD4count and viral load assessments. ART adherence and client satisfaction will be assessed at each follow-up visit while CD4count and viral load assessments will be done at baseline and at 20th week.

It is possible that tailored SMS reminders will mitigate the barrier of forgetfulness in ART-adherence and lead to improved drug compliance, viral suppression, and quality of life among adolescents living with HIV.

DETAILED DESCRIPTION:
BACKGROUND In Nigeria, approximately 3.2 million people were living with human immunodeficiency virus (HIV)/acquired immunodeficiency syndrome (AIDS) in Nigeria. Nigeria has about 196,000 adolescents (10-19 years) living with HIV with an estimated 17,000 new infections and 11,000 AIDS-related deaths per year in the age group. Adolescents aged 15 to 19 years constitute 8.8% of Nigeria's over 173 million people and have an HIV prevalence rate of 2.9%.

Non-adherence to antiretroviral therapy (ART) increases the risk of non-suppression of HIV, secondary HIV transmission, and development of drug resistance; it has a negative impact on treatment outcomes, leads to decreased survival and worsened quality of life. Adolescents on ART have lower viral suppression rates (49%) when compared with both adults and younger children (72.8% and 57%) and this is one of the most frequent causes of lower adherence to ART.

The non-maintained ART adherence is a major barrier to the achievement of optimal treatment outcomes among adolescents living with HIV. ART adherence is a challenge among adolescents living with HIV because of lack of appropriate information, their unique emotional state and lifestyles. Religious, cultural, social and health services related factors have also been recognized as a source of non-adherence to ART treatment. Other known barriers to ART adherence include difficult dosing schedule, side effects, food restrictions and pill burden but the most commonly quoted challenge to adherence is forgetting to take antiretroviral drugs. Many strategies, including directly observed drug use, adherence counselling, telephone calls and reminder devices adopted to enhance ART adherence have turned out to be time-consuming, costly and intrusive.

With over 148 million active mobile lines, short message service (SMS) has become a common means of communication in Nigeria. SMS is used commonly by teenagers, including those who are economically disadvantaged. SMS has been applied in a variety of healthcare setting because of its low-cost and convenient technology and has proved to be an effective tool for behavioural change interventions. There is evidence to suggest that SMS interventions may enhance drug compliance among adolescents living with other chronic diseases such as asthma and diabetes. An RCT showed that text-messaging system increased adherence to medication among adolescents by about 7%. While studies have evaluated the effectiveness of SMS reminders on ART adherence among PLHIV in some low-resource settings, to the best of our knowledge studies that evaluated SMS reminders for adolescents living with HIV have not yet been published. Indeed, a Cochrane systematic review of randomized controlled trials (RCTs) that assessed the effectiveness of SMS for improving ART adherence among people living with HIV infection identified the need of RCTs for this intervention among adolescents.

Mobile technology communicates interventions to people in real-time and in their natural habitat. A review of the literature on SMS interventions for behavioural change in health care settings identified key characteristics for success such as interactivity and tailored messages.

PROJECT OBJECTIVES Objective 1: To evaluate the efficacy of interactive and tailored SMS reminders on ART adherence among adolescents (15-19 years) living with HIV in Southwest, Nigeria.

Objective 2: To assess the feasibility and acceptability of using personal mobile phones and interactive and tailored SMS reminders for the improvement of ART adherence among adolescents living with HIV in Southwest, Nigeria.

Objective 3: To identify the predictors of ART non-adherence among adolescents (15-19 years) living with HIV in Southwest, Nigeria.

STUDY HYPOTHESES

1. Interactive and tailored SMS reminders are efficacious in the improvement of ART adherence among adolescents (15-19) years living with HIV.
2. The use of personal mobile phones for the improvement of ART adherence among adolescents living with HIV is feasible and acceptable.
3. ART adherence among adolescents is predicted by demographic, socioeconomic, and psychosocial factors.

METHODOLOGY Study design and procedure This study is designed to have 80% power to detect a difference of 20%. When the proportion of adolescents who are adherent to ART was taken as 49% (5), a sample size of 104 per group was obtained. The study will recruit 230 participants from the ART clinics in Southwest Nigeria into a randomized controlled trial (RCT). Convenience sampling method by which participants will be recruited on routine clinic visits across five (5) high patient-density ART sites will be used.

For the purpose of this study, we defined poor adherence as self-reported < 95% adherence in the preceding one month using a validated visual analogue scale. Self-reported 95% adherence level is an ideal cut-off point because self-reported measures tend to exaggerate adherence and such high adherence level will minimize the occurrence of false-negatives.

Initial eligibility screening and recruitment will be carried out by the primary caregivers using a checklist. Potential participants who meet the first four criteria will be presented with a visual analogue scale (VAS) labelled 0 to 100% at intervals of 5%. Eligible and willing participants will then be referred to the research assistants for a comprehensive informed consent process.

Baseline activities

At the baseline, the research assistants will give the volunteer participants a detailed explanation of the study, including its aim, duration, intervention and possible benefits. All the volunteers will be required to give a signed informed consent in a private room. Adolescents aged 15 to 19 years are thought to be relatively mature. According to a brief of AIDS regulations and Laws in Nigeria, children who are deemed mature in this context are capable of giving informed consent. Besides, based on evidence from South Africa and Lesotho, the WHO recommended that the legal age of consent for HIV testing and treatment should be 12 years. The consenting volunteers will then be allocated unique identifiers that they will maintain throughout the course of the study. The contact details of the lead investigator will be made available to the participants so that he can be reached directly for any reason that is related to the study. Baseline data will be obtained in a private room by trained research assistants using structured interviewer-administered paper-based questionnaires over a period of about 40 minutes. The questionnaire will assess:

1. socio-demographic variables.
2. HIV/AIDS risk behaviour assessment: This will be done using the AIDS Risk Behavior Assessment (ARBA); a validated, adolescent-specific tool for the assessment of sexual behaviour, drug and alcohol use, and HIV-associated needle use. It assesses sexual behaviour over the previous 30 days and the previous three months.
3. Alcohol and Drug abuse assessment: The Alcohol Use Disorders Identification Test (AUDIT) will be used to assess alcohol abuse. AUDIT, which was developed in 1982 by the World Health Organization, is a simple tool that is used to screen for and to identify people who are at risk of alcohol problems. The drug abuse screening test (DAST-20, adolescent version) will be used to screen for drug abuse. DAST is a validated scale that was designed to provide a brief, self-reported instrument for population screening, clinical case finding, and treatment evaluation research. It yields a quantitative index of the drug abuse consequences.
4. Client Satisfaction Survey: A 22-item adaptation of the SERVQUAL tool will be used for this purpose. First published in 1988, the SERVQUAL is a multi-dimensional tool that assesses patients expected and perceived quality of services across five domains. Its use currently dominates research and industry for the assessment of quality of services and is well-validated in HIV service quality assessment.
5. Adherence assessment: This will be done using the validated visual analogue scale (described above), monthly pill count, pharmacy records and the AIDS Clinical Trials Group (ACTG) adherence questionnaire. The research assistants will carry out pill counts and obtain the pharmacy records. Adherence assessment will be carried out at baseline and at every follow-up visit.

Ten millilitres (10 ml) of blood samples will also be taken by laboratory scientists to measure the volunteers' CD4 cell count and HIV viral load. Sampling collection, handling and disposal will follow the standards and guidelines outlined by the WHO and PEPFAR. The participants' capability to operate mobile phones will be enhanced. The research assistants will work with participants to select from a list the most preferred SMS that will serve as a daily reminder of ART adherence. Each participant will select an SMS format that will serve as a reminder for follow-up visit reminders. In addition, the participants will also choose the preferred language and time for SMS reminders. The messages will be designed in such a way that they are sensitive and protect the privacy of the participants. The participants will be able to contact the lead investigator if they wish to change their chosen messages or if the services to their mobile phones are disrupted.

Data Analysis The research assistants will code and enter the data obtained into Microsoft excel software in the CSV format. The data will be exported to the STATA version 15/SE for analyses. The data manager will fully review 5% (one in every twenty) questionnaire for errors. The data manager in conjunction with the investigators will be responsible for baseline, interim and final data analysis. The investigators, data manager, research assistants, counsellors and other project staff will be blinded throughout the study. After the scientific review has been completed and data collection has been completed, at the point of analysis, a list of participants' unique identifiers in two groups will be sent to the data analysts without specifying which the investigation or control group is. The blinding of the clinical database will finally be removed after final data analysis has been completed.

Statistical Methods Intention-to-treat analysis will be carried out. Baseline characteristics will be compared using the chi-square test, rank-sum test, and independent t-test as appropriate. The independent t-test will be used to compare the means of ART adherence between the investigation and control groups after each follow-up visit in order to test if the intervention has any effect. The incidence proportion, incidence rate, relative risk, risk difference, and odds ratio will be used to measure the effect. Survival analysis will also be carried out to adjust for censoring (competing risk and loss to follow-up). Multiple regression analyses will be used to control for possible confounders. Subgroup analysis will also be undertaken in order to generate further hypotheses.

The acceptability of the SMS will be accessed by the responses given by participants. The proportion of participants who find the method acceptable will be determined.

The feasibility will be determined using the proportion of participants who are deemed to have completed the study (participate fully).

The study will also assess client satisfaction and the possible effect of adherence on the mental health status of adolescents. Correlation and linear regression analyses will be used to determine the association between adherence (percent) and mental health status (GHQ 12 measure).

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositivity
* Being on ART for at least three month
* Age 15 to 19 years as at last birthday
* Use of personal mobile phone
* Poor adherence to ART

Exclusion Criteria:

Adolescents who are too ill to require hospital admission will be excluded from the study.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 212 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olumide ABIODUN, FWACP, Principal Investigator — Babcock University
Locations (5):
- Nigeria (5):
  - Lagos State University Teaching Hospital, Ikeja, Lagos
  - The Nigerian Institute of Medical Research, Yaba, Lagos
  - Federal Medical Center, Abeokuta, Ogun State
  - State Hospital, Ijebu Ode, Ogun State
  - State Hospital, Ota, Ogun State

IPD SHARING:
Plan to Share IPD: Yes
(De-identified) IPD may be shared with other researchers upon reasonable request
Supporting Information: Study Protocol
Time Frame: June 30th, 2019 to June 29th, 2020
Access Criteria: Open access Other information will be available upon reasonable request

REFERENCES:
- [Background] Dowshen N, Kuhns LM, Johnson A, Holoyda BJ, Garofalo R. Improving adherence to antiretroviral therapy for youth living with HIV/AIDS: a pilot study using personalized, interactive, daily text message reminders. J Med Internet Res. 2012 Apr 5;14(2):e51. doi: 10.2196/jmir.2015. PMID 22481246
- [Background] Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Mehendale S, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Wang L, Makhema J, Mills LA, de Bruyn G, Sanne I, Eron J, Gallant J, Havlir D, Swindells S, Ribaudo H, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano D, Essex M, Fleming TR; HPTN 052 Study Team. Prevention of HIV-1 infection with early antiretroviral therapy. N Engl J Med. 2011 Aug 11;365(6):493-505. doi: 10.1056/NEJMoa1105243. Epub 2011 Jul 18. PMID 21767103
- [Background] McMahon JH, Elliott JH, Bertagnolio S, Kubiak R, Jordan MR. Viral suppression after 12 months of antiretroviral therapy in low- and middle-income countries: a systematic review. Bull World Health Organ. 2013 May 1;91(5):377-385E. doi: 10.2471/BLT.12.112946. Epub 2013 Feb 21. PMID 23678201
- [Background] Naar-King S, Templin T, Wright K, Frey M, Parsons JT, Lam P. Psychosocial factors and medication adherence in HIV-positive youth. AIDS Patient Care STDS. 2006 Jan;20(1):44-7. doi: 10.1089/apc.2006.20.44. PMID 16426155
- [Background] Rao D, Kekwaletswe TC, Hosek S, Martinez J, Rodriguez F. Stigma and social barriers to medication adherence with urban youth living with HIV. AIDS Care. 2007 Jan;19(1):28-33. doi: 10.1080/09540120600652303. PMID 17129855
- [Background] Glikman D, Walsh L, Valkenburg J, Mangat PD, Marcinak JF. Hospital-based directly observed therapy for HIV-infected children and adolescents to assess adherence to antiretroviral medications. Pediatrics. 2007 May;119(5):e1142-8. doi: 10.1542/peds.2006-2614. Epub 2007 Apr 23. PMID 17452493
- [Background] Fjeldsoe BS, Marshall AL, Miller YD. Behavior change interventions delivered by mobile telephone short-message service. Am J Prev Med. 2009 Feb;36(2):165-73. doi: 10.1016/j.amepre.2008.09.040. PMID 19135907
- [Background] Wei J, Hollin I, Kachnowski S. A review of the use of mobile phone text messaging in clinical and healthy behaviour interventions. J Telemed Telecare. 2011;17(1):41-8. doi: 10.1258/jtt.2010.100322. Epub 2010 Nov 19. PMID 21097565
- [Background] Hung SH, Tseng HC, Tsai WH, Lin HH, Cheng JH, Chang YM. Care for Asthma via Mobile Phone (CAMP). Stud Health Technol Inform. 2007;126:137-43. PMID 17476056
- [Background] Franklin VL, Waller A, Pagliari C, Greene SA. A randomized controlled trial of Sweet Talk, a text-messaging system to support young people with diabetes. Diabet Med. 2006 Dec;23(12):1332-8. doi: 10.1111/j.1464-5491.2006.01989.x. PMID 17116184
- [Background] Miloh T, Annunziato R, Arnon R, Warshaw J, Parkar S, Suchy FJ, Iyer K, Kerkar N. Improved adherence and outcomes for pediatric liver transplant recipients by using text messaging. Pediatrics. 2009 Nov;124(5):e844-50. doi: 10.1542/peds.2009-0415. Epub 2009 Oct 12. PMID 19822583
- [Background] Lester RT, Mills EJ, Kariri A, Ritvo P, Chung M, Jack W, Habyarimana J, Karanja S, Barasa S, Nguti R, Estambale B, Ngugi E, Ball TB, Thabane L, Kimani J, Gelmon L, Ackers M, Plummer FA. The HAART cell phone adherence trial (WelTel Kenya1): a randomized controlled trial protocol. Trials. 2009 Sep 22;10:87. doi: 10.1186/1745-6215-10-87. PMID 19772596
- [Background] Horvath T, Azman H, Kennedy GE, Rutherford GW. Mobile phone text messaging for promoting adherence to antiretroviral therapy in patients with HIV infection. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD009756. doi: 10.1002/14651858.CD009756. PMID 22419345
- [Background] Heron KE, Smyth JM. Ecological momentary interventions: incorporating mobile technology into psychosocial and health behaviour treatments. Br J Health Psychol. 2010 Feb;15(Pt 1):1-39. doi: 10.1348/135910709X466063. Epub 2009 Jul 28. PMID 19646331
- [Background] Cole-Lewis H, Kershaw T. Text messaging as a tool for behavior change in disease prevention and management. Epidemiol Rev. 2010;32(1):56-69. doi: 10.1093/epirev/mxq004. Epub 2010 Mar 30. PMID 20354039
- [Background] Kalichman SC, Amaral CM, Swetzes C, Jones M, Macy R, Kalichman MO, Cherry C. A simple single-item rating scale to measure medication adherence: further evidence for convergent validity. J Int Assoc Physicians AIDS Care (Chic). 2009 Nov-Dec;8(6):367-74. doi: 10.1177/1545109709352884. PMID 19952289
- [Background] Giordano TP, Guzman D, Clark R, Charlebois ED, Bangsberg DR. Measuring adherence to antiretroviral therapy in a diverse population using a visual analogue scale. HIV Clin Trials. 2004 Mar-Apr;5(2):74-9. doi: 10.1310/JFXH-G3X2-EYM6-D6UG. PMID 15116282
- [Background] Kalichman SC, Kalichman MO, Cherry C, Swetzes C, Amaral CM, White D, Jones M, Grebler T, Eaton L. Brief behavioral self-regulation counseling for HIV treatment adherence delivered by cell phone: an initial test of concept trial. AIDS Patient Care STDS. 2011 May;25(5):303-10. doi: 10.1089/apc.2010.0367. Epub 2011 Apr 2. PMID 21457056
- [Background] Bam K, Rajbhandari RM, Karmacharya DB, Dixit SM. Strengthening adherence to Anti Retroviral Therapy (ART) monitoring and support: operation research to identify barriers and facilitators in Nepal. BMC Health Serv Res. 2015 May 5;15:188. doi: 10.1186/s12913-015-0846-8. PMID 25939593
- [Background] Watt MH, Maman S, Golin CE, Earp JA, Eng E, Bangdiwala SI, Jacobson M. Factors associated with self-reported adherence to antiretroviral therapy in a Tanzanian setting. AIDS Care. 2010 Mar;22(3):381-9. doi: 10.1080/09540120903193708. PMID 20390519
- [Background] Montazeri A, Harirchi AM, Shariati M, Garmaroudi G, Ebadi M, Fateh A. The 12-item General Health Questionnaire (GHQ-12): translation and validation study of the Iranian version. Health Qual Life Outcomes. 2003 Nov 13;1:66. doi: 10.1186/1477-7525-1-66. PMID 14614778
- [Background] Purdy JB, Freeman AF, Martin SC, Ryder C, Elliott-DeSorbo DK, Zeichner S, Hazra R. Virologic response using directly observed therapy in adolescents with HIV: an adherence tool. J Assoc Nurses AIDS Care. 2008 Mar-Apr;19(2):158-65. doi: 10.1016/j.jana.2007.08.003. PMID 18328966
- [Background] Pop-Eleches C, Thirumurthy H, Habyarimana JP, Zivin JG, Goldstein MP, de Walque D, MacKeen L, Haberer J, Kimaiyo S, Sidle J, Ngare D, Bangsberg DR. Mobile phone technologies improve adherence to antiretroviral treatment in a resource-limited setting: a randomized controlled trial of text message reminders. AIDS. 2011 Mar 27;25(6):825-34. doi: 10.1097/QAD.0b013e32834380c1. PMID 21252632
- [Background] Donenberg GR, Schwartz RM, Emerson E, Wilson HW, Bryant FB, Coleman G. Applying a cognitive-behavioral model of HIV risk to youths in psychiatric care. AIDS Educ Prev. 2005 Jun;17(3):200-16. doi: 10.1521/aeap.17.4.200.66532. PMID 16006207
- [Background] Nugent NR, Brown LK, Belzer M, Harper GW, Nachman S, Naar-King S; Adolescent Trials Network for HIV/AIDS Interventions. Youth living with HIV and problem substance use: elevated distress is associated with nonadherence and sexual risk. J Int Assoc Physicians AIDS Care (Chic). 2010 Mar-Apr;9(2):113-5. doi: 10.1177/1545109709357472. Epub 2010 Feb 4. PMID 20133498
- [Background] Shacham E, Estlund A, Presti R. Viral suppression among young adults in a US outpatient clinic. BMC Infectious Diseases 14(Suppl 2): P76, 2014. https://doi.org/10.1186/1471-2334-14-S2-P76
- [Derived] Abiodun O, Jagun O, Sodeinde K, Bamidele F, Adekunle M, David A. Socioeconomic, clinical, and behavioral characteristics of adolescents living with HIV in Southwest Nigeria: implication for preparedness for transition to adult care. AIDS Care. 2022 Mar;34(3):315-323. doi: 10.1080/09540121.2021.1906402. Epub 2021 Mar 25. PMID 33764812
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- See also: AIDSInfo for Nigeria — http://www.unaids.org/en/regionscountries/countries/nigeria
- See also: Nigeria's Phone subscribers increase to 152.1 million — http://thenewsnigeria.com.ng/2016/01/nigerias-phone-subscribers-increase-to-152-1-million/
- See also: AIDS Law Brief; Age of Consent for HIV Testing and Counseling in Nigeria — http://globalhealth.washington.edu/sites/default/files/AIDS_Law_Brief-Age_of_Consent_for_HIV%20Testing_and_Counseling_in_Nigeria.pdf
- See also: Drug Abuse Screening Test (DAST) - Adolescent Version — http://chipts.ucla.edu/wp-content/uploads/downloads/2012/02/Drug-Abuse-Screening-Test_DAST_Adolescent-Version.pdf
- See also: ACTG Adherence Baseline and Follow up Questionnaires — https://www.ghdonline.org/uploads/ACTG_Adherence_Baseline_Questionnaire.pdf
- See also: ADOLESCENT HIV TESTING, COUNSELLING AND CARE Implementation guidance for health providers and planners — http://apps.who.int/adolescent/hiv-testing-treatment/
- See also: Teens and Mobile Phones — http://www.pewinternet.org/2010/04/20/teens-and-mobile-phones/
- See also: The Alcohol Use Disorders Identification Test: Interview version — https://www.drugabuse.gov/sites/default/files/files/AUDIT.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited while attending routine clinic visits across five (5) high patient-density ART sites in 2 States in South West, Nigeria over a 13 week period.
Pre-assignment Details: There was no significant event.
Groups:
- Intervention Group: Daily ART-adherence SMS reminder
  Daily ART-adherence SMS reminder: Interactive and tailored SMS reminders that are acceptable to the participants to remind them to take their medications and to make clinic attendance.
  Standard Adherence Counselling/Patient experience group chat: All the participants will receive the standard adherence counselling by trained counsellors at each visit.
  All participants will also be enlisted in a group chat on social media where they will discuss their experiences with the quality of HIV services rendered at their respective clinics. A specialist who will have very minimal involvement will give weekly feedback and counsel on how best to resolve prominent challenges.
- Control Group: Standard adherence counselling/Patient experience group chat
  Standard Adherence Counselling/Patient experience group chat: All the participants will receive the standard adherence counselling by trained counsellors at each visit.
  All participants will also be enlisted in a group chat on social media where they will discuss their experiences with the quality of HIV services rendered at their respective clinics. A specialist who will have very minimal involvement will give weekly feedback and counsel on how best to resolve prominent challenges.
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 106 | 106
Completed | 105 | 104
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 106 | 106 | 212
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.56 (1.41) | 16.66 (1.36) | 16.61 (1.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 53 | 104
  Male | 55 | 53 | 108
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Yoruba | 67 | 67 | 134
  Hausa | 3 | 2 | 5
  Igbo | 24 | 26 | 50
  Others | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  Nigeria | 106 | 106 | 212
Baseline ART Adherence (VAS) [Count of Participants; unit: Participants] — VAS Adherence is the self-report of ART adherence using the visual analog scale. Participants reporting adherence of >/=95% have optimal adherence to the medications.
  Viral load is the number of copies of viral RNA detected in participants' blood. Participants with viral load </=20 copies per ml are regarded to have optimal viral suppression indicative of optimal adherence to medications.
  Participants
    VAS adherence (Self report of >/=95% adherence) | 0 | 0 | 0
    Viral Load </= 20 | 54 | 49 | 103

OUTCOME MEASURES:

1. Primary Outcome: ART Adherence at 20 Weeks as Determined by VAS, Viral Load
Description: ART adherence is assessed by different well-validated methods. In this study, ART adherence will be measured, primarily, using the self-report visual analog scale. The scale is well-validated, self-report of the level of ART adherence with a range from 0 to 100%. While higher values indicate better levels of adherence, patients with adherence levels of 95% and above are regarded as ART-adherent while those with values less than 95% are not adherent to ART medications.
  Viral load is the number of copies of viral RNA detected in participants' blood. Participants with viral load </=20 copies per ml are regarded to have optimal viral suppression indicative of optimal adherence to medications.
Time Frame: 20week [End of study]
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 105 | 104
Participants
  Adherence by VAS | 57 | 47
  Viral Load </= 20 copies | 63 | 46

2. Primary Outcome: ART Adherence at 20 Weeks as Determined by Pill Counts, ACTG Adherence Questionnaire, and VAS Scores
Description: AIDS Clinical Trials Group Scale scores range from 0 to 1. The higher scores reflect better ART adherence Pill count scores also range from 0 to 1 and the higher scores also reflect better adherence.
  Visual analog scale [VAS] adherence ranges between 0 and 100%. Higher scores reflect better ART adherence
Time Frame: 20week [End of study]
Measure: Mean (Standard Deviation); unit: measurement vlaues and score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 105 | 104
measurement vlaues and score on a scale
  AIDS Clinical Trials Group Scale score | 0.92 (0.15) | 0.90 (0.17)
  Pill count score score | 0.68 (0.24) | 0.65 (0.28)
  VAS score, continuous | 89.04 (11.90) | 86.99 (13.50)

3. Primary Outcome: ART Adherence at 20 Weeks as Determined by Viral Load Count
Description: Viral load count is measured in copies per ml. The minimum value is 0. There is no maximum value. The higher values reflect poor adherence
Time Frame: 20 week [End of study]
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 105 | 104
copies/mL | 11678 (51003.77) | 42676.71 (147790.6)

4. Primary Outcome: ART Adherence at 20 Weeks as Determined by Log of Viral Load Count
Description: log of viral load count is log 10 transformation of the viral load values
Time Frame: 20week [End of study]
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 105 | 104
log10 copies/mL | 1.97 (1.30) | 2.63 (1.55)

5. Secondary Outcome: Patient Satisfaction Score at 20 Weeks
Description: Patient satisfaction will be assessed using a 22-item adaptation of the SERVQUAL tool. It is a multi-dimensional service quality assessment tool that uses a 5-point likert scale scored from 1 to 5 points to assess 5 domains of client satisfaction. The domains are tangibility (4 items; scores from 4 to 20), reliability (5 items; scores from 5 to 25), responsiveness (4 items; scores from 4 to 20), assurance (4 items; scores from 4 to 20), and empathy (5 items; scores from 5 to 25). Patient satisfaction is measured by the total score which will range between 22 and 110. Higher scores indicate better client satisfaction.
Time Frame: End of Study (20weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 105 | 104
score on a scale | 88.94 (9.26) | 91.76 (8.72)

6. Secondary Outcome: Number of Participants With Mental Distress Determined by General Health Questionnaire 12 at 20 Weeks
Description: The General Health Questionnaire 12 (GHQ12) will be used to assess the mental health status of all the participants. It is a well-validated and widely used instrument for screening for mental health distress. It is a 12-item questionnaire that is based on a 4-point likert scale scored from 0 to 3 points. The scores will range between 0 and 36. A score of 12 or more is suggestive of mental distress while scores less than 12 suggest that mental distress is absent.
Time Frame: End of study (20weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 105 | 104
Participants | 2 | 11

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/106
Other Adverse Events (participants affected / at risk) | 0/106 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/91/NCT03394391/Prot_SAP_ICF_000.pdf